CLINICAL TRIAL: NCT05676073
Title: A Phase II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHEN26 Capsule in Patients With Mild to Moderate COVID-19
Brief Title: Study of SHEN26 Capsule in Patients With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Kexing Pharmaceutical Co., Ltd. (Network)
Responsible Party: Sponsor
Organization: Kexing Biopharm Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KXZY-SHEN26-101-Phase-II
Record Dates: First submitted 2023-01-03; First posted 2023-01-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHEN26 dose 1 (Experimental): SHEN26 capsule 200mg. 10 oral doses twice daily (after breakfast and dinner; Q12h±2h).
  Interventions: Drug: SHEN26 dose 1
- SHEN26 dose 2 (Experimental): SHEN26 capsule 400mg. 10 oral doses twice daily (after breakfast and dinner; Q12h±2h).
  Interventions: Drug: SHEN26 dose 2
- SHEN26 placebo (Placebo Comparator): Placebo matching the SHEN26 capsule. 10 oral doses twice daily (after breakfast and dinner; Q12h±2h).
  Interventions: Drug: SHEN26 placebo

INTERVENTIONS:
Drug: SHEN26 dose 1 — Specification: 200mg/capsule. Subjects will receive 10 oral doses twice daily (after breakfast and dinner; Q12h±2h) from Day 1 to Day 5 (or Day 1 to Day 6).
  Arms: SHEN26 dose 1
Drug: SHEN26 dose 2 — Specification: 400mg/capsule. Subjects will receive 10 oral doses twice daily (after breakfast and dinner; Q12h±2h) from Day 1 to Day 5 (or Day 1 to Day 6).
  Arms: SHEN26 dose 2
Drug: SHEN26 placebo — Placebo matching the SHEN26 capsule. Subjects will receive 10 oral doses twice daily (after breakfast and dinner; Q12h±2h) from Day 1 to Day 5 (or Day 1 to Day 6).
  Arms: SHEN26 placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-parallel-controlled phase II clinical trial. It is designed to evaluate the efficacy, safety, tolerability, and pharmacokinetic (PK) profile of SHEN26 capsules in Chinese patients with mild to moderate COVID-19.

DETAILED DESCRIPTION:
Eligible patients with mild to moderate COVID-19 will be randomized in a 1:1:1 ratio to SHEN26 low dose group (200 mg), SHEN26 high dose group (400 mg), and placebo group, with 30 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the trial's purpose, nature, methods, and possible adverse effects, volunteer as a subject, and sign the informed consent form.
2. Subjects and their female partners are willing to have no childbearing plans and voluntarily use effective contraception and have no plans to donate sperm or eggs from 2 weeks prior to screening until 6 months after the last dose of the study drug, and pledge to use one or more non-pharmacological contraceptives during sexual intercourse from 2 weeks prior to screening until 1 month after the last dose of the study drug.
3. Age 18-65 years (including boundary values, based on the time of signing the informed consent form) of either sex.
4. Positive results for SARS-CoV-2 using RT-PCR (Ct value< 25) in nasopharyngeal swab samples with the first positive nucleic acid test collected ≤ 5 days from Day 1 administration.
5. Patients with a diagnosis of mild or moderate COVID-19 at screening and/or baseline according to the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 9).
6. Liver function indicators meet the criteria of：

   * Alanine aminotransferase (ALT) ≤ 3 × ULN;
   * Aspartate aminotransferase (AST) ≤ 3 × ULN;
   * Total bilirubin (TBIL) ≤ 2 × ULN.
7. Hemoglobin (Hb) ≥ 90 g/L.
8. Platelets ≥ 100 × 10^9 /L.
9. Blood creatinine converted endogenous creatinine clearance (Ccr) > 60 mL/min (according to the Cockcroft-Gault formula).

Exclusion Criteria:

1. Subjects diagnosed with severe or critical COVID-19 at screening and/or baseline according to the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 9) or who, in the judgment of the investigator, are likely to progress to severe/critical COVID-19 prior to randomization.
2. Subjects are expected to be transferred to another hospital prior to randomization or within 72 hours of enrollment.
3. Subjects with SpO2 ≤ 93% or PaO2/FiO2 ≤ 300 mmHg, or respiratory rate ≥ 30 breaths/minute, or heart rate ≥ 125 beats/minute while breathing room air at sea level for 24 hours prior to dosing.
4. Subjects who require mechanical ventilation or are expected to require mechanical ventilation.
5. Subjects infected with COVID-19 within 3 months prior to dosing.
6. Subjects who have received SARS-CoV-2 monoclonal antibody treatment or prophylaxis within 30 days prior to dosing.
7. Subjects who have received COVID-19 convalescent plasma or COVID-19 human immunoglobulin treatment within 30 days prior to dosing.
8. Subjects who have received treatment or prophylaxis with antiviral drugs (e.g., Paxlovid, Molnupiravir, Remdesivir, lopinavir/ritonavir combination, ribavirin, chloroquine, hydroxychloroquine, etc.) within 30 days prior to dosing.
9. Subjects who have received systemic or inhaled steroids for COVID-19 treatment within 30 days prior to dosing (except for long-term stable dose treatment with concomitant chronic disease and no dose increase).
10. Subjects who are on dialysis.
11. Subjects with a history of drug or other allergies or who, in the investigator's judgment, may be allergic to the test drug or any component of the test drug.
12. Subjects who have undergone major organ surgery (excluding puncture biopsy, tracheotomy, gastrostomy, etc.) or significant trauma within 28 days prior to dosing or who require elective surgery during the trial period.
13. Subjects with a life-threatening illness within 28 days prior to dosing, or other clinically significant illness as judged by the investigator.
14. Cardiovascular disease meeting any of the following criteria:

    * Prior history of myocardial infarction within 12 months;
    * Unstable angina pectoris;
    * Clinically significant and uncontrollable cardiac arrhythmia;
    * A history of stroke or transient ischemic attack requiring medication in the past 12 months;
    * Congestive heart failure based on NYHA classification ≥ Class II;
    * Restrictive edema of ≥ grade 3 (including respiratory, chest and mediastinal disease: laryngeal edema, pulmonary edema; skin and subcutaneous tissue disease: peripheral edema);
    * Clinically uncontrollable hypertension.
15. Subjects with suspected or confirmed active systemic infections, such as bacterial, fungal, viral or other infections (other than COVID-19 infections), or with conditions that, in the investigator's judgment, would affect the assessment of endpoints in this study.
16. Subjects with known HIV infection, or human immunodeficiency virus antibody (HIV-Ab) positive at screening.
17. Subjects with liver disease meeting any of the following criteria:

    * Known active HBV infection (subjects with a history of hepatitis B or previous hepatitis B surface antigen positivity but whose liver function at baseline meets the inclusion criteria and is judged by the investigator to be stable may be enrolled);
    * Known HCV infection;
    * Primary biliary cirrhosis;
    * Child-Pugh Class B or C;
    * Acute liver failure.
18. Subjects who have difficulty with venous blood collection or have a history of acupuncture and blood sickness.
19. Female subjects who have tested positive for pregnancy or are breastfeeding during the screening or baseline period.
20. Subjects who have participated in other drug clinical trials and used other clinical trial drugs within 1 month prior to screening.
21. Subjects who have received any vaccine within 1 month prior to screening or subjects who are scheduled to receive vaccines (including COVID-19 vaccine boosters) during the trial.
22. Any other circumstances that, in the investigator's opinion, may affect the subject's ability to provide informed consent or follow the trial protocol, or the subject's participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 viral RNA level (RT-PCR) on Day 7 | Day 7
  Change from baseline in SARS-CoV-2 viral RNA level (RT-PCR) on Day 7

SECONDARY OUTCOMES:
TEAEs and SAEs | From Baseline up to Day 28
  The incidence of treatment-emergent adverse events (TEAE) and serious adverse events (SAEs).
AEs leading to discontinuation of treatment | From Baseline up to Day 28
  The incidence of AEs leading to discontinuation of study treatment.
Drug-related treatment discontinuation | From Baseline up to Day 28
  The incidence of drug-related study treatment discontinuation.
New AEs of Grade 3 or higher | From Baseline up to Day 28
  The incidence of new Grade 3 or higher AE (not present at baseline).
  The investigator should classify the severity of adverse events (AEs) into Grades 1 to 5 according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, with Grade 1 being the least severe and Grade 5 the most.
New drug-related AEs of Grade 3 or higher | From Baseline up to Day 28
  Incidence of new drug-related AEs of Grade 3 or higher.
  The investigator should classify the severity of adverse events (AEs) into Grades 1 to 5 according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, with Grade 1 being the least severe and Grade 5 the most.
SARS-CoV-2 viral RNA level (RT-PCR) at prespecified timepoints | Day 3, Day 5, Day 7, Day 10, Day 28
  Change from baseline in SARS-CoV-2 viral RNA level (RT-PCR)
Time to achieve SARS-CoV-2 viral clearance | From Baseline up to Day 28
  Viral clearance is defined as two consecutive viral nucleic acid assays with Ct values ≥35 for both N and ORF genes by RT-PCR and an interval of ≥24 hours between sampling. The date of achieving clearance is calculated as the date of the first Ct value ≥ 35).
Percentage of participants achieving SARS-CoV-2 viral clearance at prespecified timepoints | Day 3, Day 5, Day 7, Day 10, Day 28
  The change in percentage of participants achieving SARS-CoV-2 viral clearance.
Plasma concentrations of SHEN26-69-0 on Day 5 | Day 5
Time to achieve sustained alleviation of COVID-19 symptoms | From Day 1 up to Day 28
  Time to achieve sustained alleviation of 11 symptoms of COVID-19 after the first dose, with sustained alleviation defined as a related symptom score of 0 to 1 and lasting ≥ 48 hours.
  The severity of symptoms will be scored according to the COVID-19 Major Symptoms and Rating Scale, with 0 being the least severe and 3 being the most.
Time to achieve sustained recovery of COVID-19 symptoms | From Day 1 up to Day 28
  Time to achieve sustained recovery of 11 symptoms of COVID-19 after the first dose, with sustained recovery defined as a relevant symptom score of 0 and lasting ≥ 48 hours.
  The severity of symptoms will be scored according to the COVID-19 Major Symptoms and Rating Scale, with 0 being the least severe and 3 being the most.

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, MD, PhD, Principal Investigator — Shenzhen Third People's Hospital
Locations (4):
- China (4):
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - The Third People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Shenzhen Longhua District People's Hospital, Shenzhen, Guangdong
  - Shijiazhuang Fifth Hospital, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bai J, Asakawa T, Yuan W, Lin Y, Ju H, Xu D, Yang M, Li S, Li G, Guo D, Lu H, Zhang X. Efficacy and safety of SHEN26, a novel oral small molecular RdRp inhibitor for COVID-19 treatment: a multicenter, randomized, double-blinded, placebo-controlled, phase II clinical trial. Virol J. 2025 Jan 25;22(1):16. doi: 10.1186/s12985-025-02631-y. PMID 39863888